CLINICAL TRIAL: NCT01893203
Title: Treatment of AKs With Daylight-PDT: Comparing Two Photosensitizers (BF-200 ALA and MAL)
Brief Title: Daylight-PDT for AKs: Comparing Two Photosensitizers (BF-200 ALA and MAL)
Acronym: 2013-002108-15
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R13073 / Q257; 2013-002108-15 (EudraCT Number)
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Actinic Keratoses
MeSH Terms: interventions — Aminolevulinic Acid; methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BF-200 ALA vs MAL (Other): BF-200 ALA cream and MAL (Metvix, Galderma) used in a randomized split-face design
  Interventions: Drug: BF-200 ALA cream; Drug: MAL cream

INTERVENTIONS:
Drug: BF-200 ALA cream — The symmetrical treatment areas will be randomized for treatments. First the treatment area will be wiped ethanol. Then sun protection factor (SPF) 20 cream will be applied on all sun-exposed areas of the skin. Then a 0,25mm layer application of Ameluz cream on the area. After appropriate absorption time of 30 minutes, the patients will be taken to the hospital balcony for 2 hour illumination with daylight to accomplish the phototoxic reaction. Maximum dosage will be 2 grams. The treatment will be repeated after 2 weeks for thicker gr II-III lesions with the same protocol.
  Other Names: 5-aminolaevulenic acid nanoemulsion; Ameluz
Drug: MAL cream — The symmetrical treatment areas will be randomized for treatments. First the treatment area will be wiped ethanol. Then SPF20 sun protection cream will be applied on all sun-exposed areas of the skin. Then a 0,25mm layer application of Metvix cream on the area. After appropriate absorption time of 30 minutes, the patientswill be taken to the hospital balcony for 2 hour illumination with daylight to accomplish the phototoxic reaction. Maximum dosage will be 2 grams. The treatment will be repeated after 2 weeks for thicker gr II-III lesions with the same protocol.
  Other Names: methylaminolevulinic acid; Metvix

SUMMARY:
The aim of the study is to compare the efficacy of two photosensitizers, methyl-aminolaevulinate (MAL) and 5-aminolaevulinic nanoemulsion (BF-200 ALA) in the treatment of facial actinic keratosis. We use randomized, double-blinded prospective study design. The efficacy will be assessed clinically, histopathologically and immunohistochemically.

DETAILED DESCRIPTION:
Actinic keratoses (AKs) are superficial premalignant skin lesions that can progress into an invasive or metastatic squamous cell carcinoma. AKs can be treated with photodynamic therapy (PDT), of which cure rate compares to cryo surgery with an excellent cosmesis. In PDT the AK lesions are first curettaged, then a photosensitizer is applied on the skin and let to absorb for 3 hours. The skin is illuminated using a blue or red light source light source depending on the photosensitizer, which induces activation of protoporphyrin IX (PpIX) and phototoxic reaction destroying the cancer cells.

The approved photosensitizers in Europe are methyl-aminolevulinic acid cream, (MAL, Metvix™, Galderma), a patch containing 5-aminolevulinic acid (5-ALA, Alacare®, Spirig AG) and 5-aminolevulinic acid gel (BF-200 ALA, Ameluz®, Biofrontera AG) to be used with a red LED light (630-635 nm). In North America a 5-aminolevulinic acid stick (5-ALA, Levulan® Kerastick) can also be used with a blue light source (417 nm).

PpIX absorption peaks are within the visual spectrum of light, which allows PpIX daylight activation. During natural daylight PDT (NDL-PDT) protocol, PpIX is continuously activated during its development, whereas in conventional PDT (LED-PDT) using red LED lamps, large amounts of accumulated PpIX are momentarily activated.

Since skin field cancerization refers to presence of different degrees of visible and invisible dysplastic changes, the whole area should be treated to prevent the development of non-melanoma skin cancers (NMSCs). NDL-PDT enables treatment of field cancerization in one sitting whereas LED-PDT may need repeated illuminations to cover the whole area. NDL-PDT results in enhanced cost-efficacy due to reduced staff expenses, since there's no need for sensitizer absorption and illumination.

At the moment two photosensitizers have marketing authorization in Finland, ALA (Ameluz®) and MAL (Metvix™). We are piloting a study comparing the efficacy of these two light sensitizers in NDL-PDT. The efficacy of the treatments will be assessed clinically, histopathologically and immunohistochemically.

ELIGIBILITY:
Inclusion Criteria:

* actinic keratoses symmetrically on face or scalp
* age over 18 years
* there must be at minumum one ak sized 6mm2 symmetrically on both sides
* patients must be able to make the decision to attend independently

Exclusion Criteria:

* pregnancy
* lactation
* lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noora E Neittaanmäki-Perttu, MD, Principal Investigator — Helsinki University Central Hospital; Toni T Karppinen, MD, Principal Investigator — Päijät Häme Central Hospital; Taneli Tani, PhD, Study Chair — Päijät Häme Central Hospital
Locations (1):
- Päijät-Häme Central Hospital, Lahti, Finland

REFERENCES:
- Available data/document: Clinical Study Report: 25109244 — http://www.ncbi.nlm.nih.gov/pubmed/

RESULTS

PARTICIPANT FLOW:
Groups:
- BF200 ALA vs MAL: 5-aminulevulinic acid nanoemulsion (BF-200 ALA, Ameluz, Biofrontera) and methylaminolevulinic acid (MAL, Metvix, Galderma) in randomized split face design on symmetrical treatment areas.
Period: Overall Study
Arm/Group | BF200 ALA vs MAL
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 14 patients were recruited. One withdrew because of conditions not related to the study. This patient was not included in the analysis.
Arm/Group | BF-200 ALA vs MAL
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 79.8 [66 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Number of AKs [Number; unit: Number of actinic keratoses (AKs)] | 177

OUTCOME MEASURES:

1. Primary Outcome: Histological Lesion Clearance
Description: Punch biopsies were taken symmetrically on both treatment fields from equally graded >6 mm AKs prior to treatment and again at 3 months, blinded observer (pathologist). HE- and p53-stainings. Samples not fulfilling the criteria of an AK were defined as healthy or completely cleared. The p53 reactivity expressed as average percentage of positive nuclei in three consecutive high power fields from the region of highest reactivity (<10 % normal)
Time Frame: 0 (baseline) and 3 months
Population: Punch biopsies bilaterally on treatment fields
Measure: Number; unit: percentage of complete clearance
Groups:
- BF200 ALA vs MAL: BF-200 ALA (Ameluz, Biofrontera) and MAL (Metvix, Galderma) in randomized split face design on symmetrical treatment areas.
Arm/Group | BF200 ALA vs MAL
Number analyzed (Participants) | 13
percentage of complete clearance
  BF-200 ALA | 61.5
  MAL | 38.5
Statistical Analysis 1: Comparison: BF200 ALA vs MAL; Test type: Superiority or Other; p = 0.375, McNemar

2. Secondary Outcome: Pain
Description: Pain using visual analog scale (VAS 0-10, where 0 is no pain and 10 is the worst pain imaginable) on both treatment sides is assessed in every 30 minutes during 2-hour sun-exposure and afterwards once in two hours until 9 p.m.
  (treatment day). Of these values, the mean maximal pain is assessed.
Time Frame: 12 hours
Population: Patients
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BF200 ALA vs MAL
Number analyzed (Participants) | 13
units on a scale
  BF-200 ALA treatment sides | 1.7 [0.4 to 8.6]
  MAL treatment sides | 1.9 [0.2 to 8.6]

3. Secondary Outcome: Clinical Lesion Clearance
Description: Clinical lesion clearance is observed by a blinded observer
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of complete clearance
Units Other Than Participants: AKs total
Arm/Group | BF200 ALA vs MAL
Number analyzed (Participants) | 13
Number analyzed (AKs total) | 177
percentage of complete clearance
  BF-200 ALA treated lesions | 84.5 [75.2 to 90.9]
  MAL treated lesions | 74.2 [64.4 to 82.1]

4. Other Pre Specified Outcome: Adverse Reactions
Description: Adverse reactions are evaluated by blinded observer at one week after treatment. A dermatologist will assess which side of the face or scalp presents a stronger reaction.
Time Frame: 1 week
Population: One week after the first photodynamic therapy (PDT), seven patients had more severe reactions (erythema, crusting) at the site treated with BF-200 ALA, five patients had more severe reactions at the MAL site and one patient showed no difference between sites.
Measure: Number; unit: participants
Arm/Group | BF200 ALA vs MAL
Number analyzed (Participants) | 13
participants
  BF-200 ALA treated areas | 7
  MAL treated areas | 5
  No difference between the sides | 1

ADVERSE EVENTS:
Groups:
- BF200 ALA vs MAL: BF-200 ALA (Ameluz, Biofrontera) and MAL (Metvix, Galderma) in randomized slipt face design on symmetrical treatment areas.
Arm/Group | BF200 ALA vs MAL
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF200 ALA vs MAL (N=13)
Adverse reactions: erythema, crusting, scaling (Skin and subcutaneous tissue disorders) | 13 (13) — Erythema, crusting and scaling were assessed all together as one score of mild, moderate or severe
Pain (Skin and subcutaneous tissue disorders) | 13 (13) — Pain in VAS scale 1-10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No